CLINICAL TRIAL: NCT02323932
Title: Perception of Intonation by Bimodal and Bilateral Cochlear Implant Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, MICHAL.LUNTZ, Head of Otolaryngology Head and Neck Department, Bnai Zion Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BZ0085
Record Dates: First submitted 2014-12-15; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilateral Cochlear implant users (Active Comparator): The perception of intonation will be assessed through the use of 2 tests. In the first test, listeners will have to identify statements and yes/no questions that will be presented by male and female talkers in the background of four- talkers-babble noise comprised of two females and two males. In the second test, listeners will be presented with gradual changes in the fundamental frequency of a sentence. They will be required to identify the sentence with each of the changes as a statement or a question. Each of the 2 tests will be presented in three listening conditions: each of the CI alone and bilateral (CI/CI) conditions.
  Interventions: Behavioral: Perception of correct intonation identification
- Bimodal Cochlear implant users (Active Comparator): The perception of intonation will be assessed through the use of 2 tests. In the first test, listeners will have to identify statements and yes/no questions that will be presented by male and female talkers in the background of four- talkers-babble noise comprised of two females and two males. In the second test, listeners will be presented with gradual changes in the fundamental frequency of a sentence. They will be required to identify the sentence with each of the changes as a statement or a question. Each of the 2 tests will be presented in three listening conditions: CI alone, HA alone and bimodal (CI/HA) conditions.
  Interventions: Behavioral: Perception of correct intonation identification

INTERVENTIONS:
Behavioral: Perception of correct intonation identification — The amount of change in the fundamental frequency that was required in order to identify a question

SUMMARY:
The purpose of this study is to evaluate the benefit of bimodal hearing and bilateral cochlear implant hearing in comparison to unilateral cochlear implant hearing in the perception of speech intonation.

DETAILED DESCRIPTION:
Bilateral hearing which is a fundamental characteristic of normal auditory system provides significant advantages in adverse listening conditions. In cochlear implant users, binaural hearing can be achieved via bilateral cochlear implant (CI/CI) or binaural-bimodal stimulation, i.e. a cochlear implant in one ear and a hearing aid in the other (CI/HA). It is assumed that CI/CI hearing and CI/HA hearing differ with respect to their physiological sources and functional benefit. Although both hearing prosthesis (CI/CI or CI/HA) lack several of the features needed to allow listeners to experience the full binaural advantage conferred by a normal-hearing auditory system it can, however, provide significant advantages over the use of a unilateral hearing prosthesis. Most of the accepted assessment clinical materials are not sensitive enough to evaluate the contribution of binaural hearing rehabilitation via CI/CI or CI/HA hearing for the perception of intonation. In a previous study the perception of intonation was evaluated in 29 adults CI/HA users via a closed-set format design with the same target talker. The results of the study showed small bimodal benefit. The test paradigm was apparently an easy task for the adult listeners and not sensitive enough to show the expected CI/HA bimodal benefit over cochlear implant alone.

The perception of correct intonation identification will be computed for each listener in each of the listening conditions. The amount of change in the fundamental frequency that was required in order to identify a question will be computed for each listener in each of the conditions. ANOVA with repeated measures will be used to assess the differences among the conditions for each group as well as the differences among the groups.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cochlear implant users
* Bilateral-bimodal users who use hearing aids for at least 75% of their waking hours.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The amount of change in the fundamental frequency that was required in order to identify a question | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michal Luntz, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnzi Zion Medical Center, Haifa, Israel